CLINICAL TRIAL: NCT05484830
Title: Impact of Anticoagulation Management on Thrombin Generation During Surgery for Acute Aortic Dissection
Brief Title: Coagulation in Acute Aortic Dissection
Acronym: CAAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivy susanne Modrau, MD (Other)
Responsible Party: Sponsor-Investigator, Ivy susanne Modrau, MD, Dr. Med., Consultant Cardiac Surgeon, Associate Professor, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-30-22
Record Dates: First submitted 2022-05-26; First posted 2022-08-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Acute Aortic Dissection; Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Investigator-initiated single-site paralle-group (1:1) prospective, randomized, partially double-blinded trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Treatment group allocation cannot be concealed for the operating team, but participants, other members of the treatment team, laboratory personnel and other practitioners administering postoperative care as well as outcome assessors will be blinded regarding the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualised HDR-approach (Active Comparator): HMS Plus® Hemostasis Management System (Medtronic International, Tolochenaz, CH).
  Interventions: Procedure: Individualized HDR-approach
- Conventional ACT-approach (Active Comparator): ACT Hemostasis Management
  Interventions: Procedure: Conventional ACT-approach

INTERVENTIONS:
Procedure: Individualized HDR-approach — Heparin concentration necessary to achieve target ACT > 480 sec. calculated based on individual HDR-curve.
  If HDR slope ˂80 s/IU/mL (reduced sensitivity to heparin), 1000 IU of AT concentrate (Antitrombin III "Baxalta"®, Takeda Pharma, Vallensbæk Strand, DK). Whole blood concentration of circulating heparin assessed by heparin assays. Additional heparin given as required. After weaning, protamine necessary to reverse circulating heparin calculated according to heparin-protamine titration measurement. After protamine, heparin reversal evaluated with low-range heparin-protamine titration cartridge and additional protamine given as required.
  Arms: Individualised HDR-approach
Procedure: Conventional ACT-approach — Initial Heparin 400 IU/kg (500 IU/kg if treated with heparin prior to surgery). ACT Assessment with Hemochron® Signature Elite (ITC, International Technidyne Corp., Edison, NJ, USA).
  Additional heparin until ACT > 480 sec. If ACT < 480 sec. after despite repeated heparin supplement with 1000 IU of AT III concentrate. Target ACT > 480 sec. during normothermic CPB, and target ACT > 700 seconds during hypothermia After weaning, protamine 10mg/mL (0.7 mg of protamine/ 100 IU total heparin administered). Heparin reversal is evaluated with an activated partial thromboplastin (APTT). If APTT > 40 seconds, additional protamine (25-50 mg i.v.).
  Arms: Conventional ACT-approach

SUMMARY:
Acute aortic dissection (AAD) involving the ascending aorta (Stanford classification type A) remains a life-threatening disease. Excessive perioperative bleeding requiring massive transfusion of allogeneic blood products, and surgical reexploration remain major challenges in these patients. Previous research has indicated that patients with AAD show pronounced haemostatic alterations prior to surgery which are aggravated during major aortic surgery with cardiopulmonary bypass and hypothermia full heparinization.

Intensified anticoagulation management guided by heparin dose response (HDR) calculation, and repeated measurement of heparin concentration may be more effective than standard empiric weight-based heparin and protamine management monitored by activated clotting time (ACT) measurements to suppress thrombin generation during surgery for AAD.

This randomized controlled clinical trial compares the impact of two recommended anticoagulation management strategies during surgery for AAD including deep hypothermia on activation of coagulation: Heparin/protamine-management based on HDR-titration by means of HMS Plus® versus current institutional standard (HDR- versus ACT-approach).

Primary endpoint is thrombin generation as measured by early postoperative prothrombin fragment 1+2 (F1+2). Secondary endpoints are other markers of coagulation and fibrinolysis as well as clinical outcome.

DETAILED DESCRIPTION:
Hypotheses:

Primary: HDR-approach is superior to ACT-approach in terms of suppressing thrombin generation after emergent surgery for acute aortic dissection (Stanford type A).

Secondary: HDR-approach is superior with regard to

* early postoperative haemostatic capacity
* requirement of blood product transfusion and haemostatic agents
* postoperative bleeding

Design:

Investigator-initiated, single-site, parallel-group (1:1), prospective, randomized, partially double-blinded trial in patients undergoing emergent surgery for acute aortic dissection comparing two heparin management strategies with superiority design. Prior to randomization, patients are stratified according to preoperative organ dysfunction and anticoagulation therapy.

Acute research study design as patients with acute aortic dissection are considered incompetent according to the Danish Research Ethics Committees definition. Deferred consent by the competent patient or her/his proxy (next of kin) and an independent physician) is used. 26 consecutive patients undergoing emergent surgery for acute aortic dissection (Stanford type A) are randomized 1:1 into the following heparin management strategies with an ACT target of 480 seconds:

* Individualised HDR-approach
* Conventional ACT-approach

No interim analysis. A sub-study to compare cost-benefit of both strategies is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Emergent Acute Aortic Dissection with cardiopulmonary bypass
* Incapable of providing informed consent

Exclusion Criteria:

* History of congenital coagulation disorder (haemophilia)
* Previous open cardiac surgery
* Death during induction of anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
F1+2 | up to 2 days after surgery
  Prothrombin fragment 1+2 (pmol/L)

SECONDARY OUTCOMES:
TAT | up to 2 days after surgery
  Thrombin-Antithrombin Complex (ug/L)
ETP | up to 2 days after surgery
  Endogenous Thrombin Potential (nmol/L x min)
Thrombin time | up to 2 days after surgery
  High-dose thrombin time (sec)
Antithrombin | up to 2 days after surgery
  (kIU/L)
D-dimer | up to 2 days after surgery
  D-dimer (mg/L)
Clot lysis | up to 2 days after surgery
  Clot lysis
Heparin sensitivity | prior to surgery
  Heparin sensitivity (slope)
Heparin (total) | immediately after surgery
  Total amount of heparin
Protamin (total) | immediately after surgery
  Total amount of protamin
Ratio | immediately after surgery
  Protamin/heparin ratio
Resistance | immediately after surgery
  Heparin resistance
Blood cell-saver | immediately after surgery
  Volume of blood processed in cell-saver (mL)
Blood loss sponges | immediately after surgery
  Gravimetric estimation of intraoperative blood loss (calculation based on the change between dry and blood-soaked sponges, accounting for irrigation) in mL
Drain output | 48 hours after surgery
  Total mediastinal drain output (ml)
Blood tranfusion | 48 hours after surgery
  Tranfusion of blood products (units): Red blood cells, fresh frozen plasma, platelet concentrates
Fibrinogen | 24 hours after surgery
  Administration of fibrinogen concentrate (mg)
PCC | 24 hours after surgery
  Administration of prothrombin complex concentrate (Octaplex) (IU)
AT concentrate | 24 hours after surgery
  Administration of Antithrombin concentrate (IU)
Cryoprecipitate Plasma | 24 hours after surgery
  Administration of cryoprecipitate plasma
Recombinant FVIIa | 24 hours after surgery
  Administration of Recombinant FVIIa
2. Closure | 30 days after surgery
  Secondary closure
Reoperation for bleeding | 30 days after surgery
  Reexploration for bleeding (yes/no)
Protocol violation | immediately after surgery
  Protocol violation (yes/no)
Mortality | up to 90 days after surgery
  All-cause mortality
Stroke | 30 days after surgery
  Stroke (yes/no)
Myocardial infarction | 30 days after surgery
  Perioperative myocardial infarction (yes/no)
Renal | 30 days after surgery
  Requirement of continuous renal replacement therapy (yes/no)
Low cardiac output syndrome | 30 days after surgery
  Low cardiac output syndrome requiring inotropics or mechanical support (yes/no)
Vascular malperfusion | 30 days after surgery
  Visceral og peripheral vascular malperfusion requiring surgical or percutaneous intervention
Intraop. coagulation | Immediately after surgery
  Clinical signs of coagulation during CPB (yes/no)
Length of surgery | 30 days after surgery
  minutes
Length of stay ICU | 30 days after surgery
  days
Length of hospitalization | 30 days after surgery
  Hospitalization (days)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eschen, Stud.med., Principal Investigator — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Denmark; Ivy Modrau, MD, dr.med., Study Chair — University of Aarhus
Locations (1):
- Aarhus University Hospital Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No